CLINICAL TRIAL: NCT04629872
Title: Combinating Fingolimod With Endovascular Treatment in Acute Ischemic Stroke
Brief Title: Fingolimod in Endovascular Treatment of Ischemic Stroke
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ning Wang, MD., PhD. (Other)
Responsible Party: Sponsor-Investigator, Ning Wang, MD., PhD., Director of Neurology department, First Affiliated Hospital of Fujian Medical University
Organization: First Affiliated Hospital of Fujian Medical University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MRCTA, ECFAH of FMU [2020]296
Record Dates: First submitted 2020-11-11; First posted 2020-11-16 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Stroke Inflammation
MeSH Terms: interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- endovascular treatment with fingolimod (Experimental)
  Interventions: Drug: Fingolimod
- endovascular treatment without fingolimod (No Intervention)

INTERVENTIONS:
Drug: Fingolimod — Patients randomized to fingolimod will also receive oral fingolimod (Gilenya, Novartis) at a dosage of 0.5 mg once daily, for three consecutive days, with the first dose being given at the time in which patients are enrolled which is more than 3 hour prior to mechanical thrombectomy.
  Arms: endovascular treatment with fingolimod

SUMMARY:
Proof-of concept clinical trials have indicated that the sphingosine-1-phosphate receptor modulator fingolimod may be efficacious in attenuating brain inflammation and improving clinical outcomes in patients with acute ischemic stroke as a single therapy beyond 4.5 hours of disease onset, or in combination with alteplase within 4.5 hours of disease onset. This study aim to determine whether fingolimod enhance the action of endovascular treatment for acute ischemic stroke

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with anterior circulation acute ischaemic stroke who are eligible for mechanical thrombectomy commenced within 6-24 hours of stroke onset.
* Patient, family member or legally responsible person depending on local ethics requirements has given informed consent.
* Patient's age is 18-80 years.
* Arterial occlusion on internal carotid artery proximal or middle cerebral artery
* Imaging inclusion criteria: infarct core volume between 15-70 mL

Exclusion Criteria:

* Pre-existing neurologic disability (a score greater than 2 on the mRS).
* Swallowing difficulties that would prevent administration of oral fingolimod.
* Patients with any history of bradyarrhythmia, atrioventricular block or current use of beta-blockers or verapamil.
* Patients with serious acute or chronic infection, or hepatic injury
* Concomitant use of antineoplastic, immunosuppressive or immune modulating therapies.
* Macular edema.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-11-12 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
the grade of collateral circulation | Baseline (before endovascular treatment)
  Multiphasic contrast-enhanced CT collateral grades with six-point pial arterial filling ordinary score as established at the University of Calgary

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Fujian Medical University, Fuzhou, China

IPD SHARING:
Plan to Share IPD: No